CLINICAL TRIAL: NCT04667689
Title: Phase II SBIR - CAMPFIRE: An Electronic Platform for Cognitive Assessment in Cancer Patients
Brief Title: An Online Cognitive Assessment in Cancer Patients
Acronym: CAMPFIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Charles River Analytics (Industry)
Responsible Party: Principal Investigator, Michelle Janelsins, PhD, MPH, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS19151
Record Dates: First submitted 2020-11-12; First posted 2020-12-16 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Cancer-Related Cognitive Difficulties; Cancer-Related Cognitive Impairment
Keywords: Cancer; Cognition
MeSH Terms: conditions — Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAMPFIRE Assessment (Other): NIH Toolbox Cognitive Assessment and PROMIS Surveys
  Interventions: Behavioral: CAMPFIRE Online Cognitive Assessment for Cancer Patients

INTERVENTIONS:
Behavioral: CAMPFIRE Online Cognitive Assessment for Cancer Patients — Subjects will complete PROMIS Cognitive Function/Anxiety/Depression survey assessments and a short neuropsychological battery (NIH Toolbox) on an iPad while in clinic prior to beginning chemotherapy, again before a clinic visit scheduled between 6 - 9 weeks and, lastly, before a post-chemotherapy follow-up clinic visit. Within two weeks of their post-chemotherapy assessment, subjects will be asked to complete a feedback survey. The physician providers and/or their clinical team (e.g., nurse practitioners, registered nurses) will be asked to review subjects' cognitive assessment results and discuss referrals and/or recommendations, if appropriate.
  Other Names: CAMPFIRE (Cognitive Assessment and Monitoring Platform for Integrative Research) system

SUMMARY:
The purpose of this study is to test the feasibility (acceptability and usability) and usefulness of the CAMPFIRE (Cognitive Assessment and Monitoring Platform for Integrative Research) system, a patient-facing portal able to collect and produce reports for clinicians on Patient Reported Outcome Measurement Information System (PROMIS-Cognitive Function/Anxiety/Depression) outcomes via MyChart and NIH Toolbox, an inperson brief objective cognitive function battery. This study will aim to determine the value of the CAMPFIRE system for patients and providers as a tool for monitoring cognitive symptoms throughout the course of chemotherapy

DETAILED DESCRIPTION:
CAMPFIRE is a health informatics platform and research tool that seeks to improve clinical research and treatment of cognitive sequelae of cancer and chemotherapy. CAMPFIRE provides curated digital assessments with content specifically for cognitive and psychosocial function assessment, and automates and integrates the data collection, analysis and visualization process into clinical workflows. CAMPFIRE is designed to both improve the availability of data on cognitive impairments among cancer patients, and to improve the integration of the produced data into the care process to efficiently improve outcomes. Key to the overall success of CAMPFIRE is the inclusion of well-validated measures to assess function in cognitive domains often affected in cancer patients, including attention, executive function, working memory, verbal and visuospatial abilities and verbal fluency.

The subjects will be asked to complete a cognitive assessment survey through a link to CAMPFIRE PROMIS in their MyChart account prior to beginning chemotherapy, between 6 - 9 weeks and prior to a post-chemotherapy follow up clinic visit. Subjects will also be asked to complete a brief cognitive assessment (NIH Toolbox) on an iPad in the JPWCI prior to their scheduled clinic visits at the same three study assessment time points.

ELIGIBILITY:
Inclusion Criteria:

* Must have diagnosis of cancer
* Must be scheduled to receive any standard course of curative intent cytotoxic chemotherapy
* Must have a computer, a general knowledge of how to use a computer and access to the internet
* Must be able to speak and read English
* Must be 21 years or older
* Must provide informed consent

Exclusion Criteria:

* Must not be currently hospitalized or have been hospitalized for any psychiatric illness within the last year
* Must not be diagnosed with neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease)
* Must not have any CNS disease (e.g., movement disorder, multiple sclerosis)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Completion | Post-Chemotherapy (16-18 weeks)
  To determine the proportion of patients who complete the full-scope CAMPFIRE NIH PROMIS and NIH Toolbox battery throughout treatment (i.e., pre-chemotherapy time-point, 6-9 week time-point, post-chemotherapy time-point) Among the enrolled patients we will calculate proportions of patients who complete the full CAMPFIRE workflow at multiple time points: (1) at pre-chemotherapy; (2) at post-chemotherapy; and (3) at any time point in between. Similarly, proportions of completers will be calculated for each collection of measures for CAMPFIRE (NIH PROMIS and NIH Toolbox). The differences in completion of tests by age and gender will be compared. For individual tests, we will determine the proportion of patients completing the test and use descriptive statistics to summarize data. Descriptive statistics will be used to characterize the cohort of enrolled patients.

SECONDARY OUTCOMES:
Provider Action | Post-Chemotherapy (16-18 weeks)
  To determine the proportion of patients for which the providers read and make any action (e.g., note in medical record, follow-up referral and types of follow-up referrals) based on the study assessments.
  For each provider and time point, we will evaluate the number (and proportion) of patients for whom: (1) the provider read the assessment and made any type of note; and (2) the provider determined particular follow-up actions. We will evaluate the differences among providers and also the differences from pre- to post-chemotherapy for the same provider. We will describe the patterns of the type of follow-up action, if any, using quantitative analysis of referrals. It will be recorded if and when providers conduct any follow-up action, up to one month post-chemotherapy.
  A Provider Behaviors Form will be completed by the study coordinator at each time-point to record information about CAMPFIRE data and how and when the provider responded to it.
Changes in Cognition via NIH Toolbox Assessment | Post-Chemotherapy (16-18 weeks)
  To assess longitudinal changes in cognition from pre-treatment through follow-up using NIH Toolbox assessment tools. The assessment of cognition will include the following two NIH Toolbox tests: Picture Sequence Memory Test and and Flanker Inhibitory Control and Attention Test.
  All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 6-9 week and post-chemotherapy time-points to baseline with t-tests and ANCOVAs adjusting for relevant covariates including age, sex, cancer type, chemotherapy regimen, and depression and anxiety scores. Additionally we will conduct linear mixed model analysis incorporating together data from all 3 time points.
Changes in Cognition via PROMIS Surveys | Post-Chemotherapy (16-18 weeks)
  To assess longitudinal changes in cognition from pre-treatment through follow-up using NIH Toolbox assessment tools. The assessment of cognition will also include the PROMIS-Cognitive Function/Anxiety/Depression surveys. The PROMIS survey assessment scores will include subject's overall perceived symptom score, how it compares to the population median, and the results of 8 subdomains.
  All cognitive data will be represented by raw scores and T scores. We will assess changes over time in patients comparing their 6-9 week and post-chemotherapy time-points to baseline with t-tests and ANCOVAs adjusting for relevant covariates including age, sex, cancer type, chemotherapy regimen, and depression and anxiety scores. Additionally we will conduct linear mixed model analysis incorporating together data from all 3 time points.
Participant Feedback | Post-Study (18-20 weeks)
  To qualitatively assess patient and provider feedback about the preferences for cognitive data type (self-report, objective) and workflow (timing of assessments, delivery methods of data).
  Participants will complete a Feedback Survey within two weeks following their completion of the Post-Chemo assessment. Provider participants will complete a Feedback Survey at the time the first participant under their care completes the Post-Chemo assessment.
  We will summarize the data from patients' and physicians' feedback forms, using frequencies and descriptive statistics. Feedback collected from participants and provider participants will be integrated and analyzed together. The focus will be on detecting systematic procedures in the CAMPFIRE application (e.g., flow) and cognitive assessment measures and outcome data presentation that work well and could be improved in order to inform the design of the future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Janelsins, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States